CLINICAL TRIAL: NCT01523665
Title: Evaluation of Blood Glucose Control in Intensive Care Patients Using the Space GlucoseControl System
Brief Title: Blood Glucose Control in Intensive Care Patients Using the Space GlucoseControl System
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HC-O-H-1102
Record Dates: First submitted 2012-01-26; First posted 2012-02-01 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Intensive Care Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Glucose metabolism is impaired in many critically ill patients and is often aggravated by parenteral feeding, infections and/or pre-existent diabetes.Therefore insulin infusion protocols, which are based on frequent bedside glucose monitoring, have been implemented on most critical care units. Despite extensive efforts of the intensive care unit staff difficulties were experienced in achieving efficient and safe glucose control. Several barriers to the implementation of glycemic control have been identified. Most importantly, there is concern about increased frequency of severe hypoglycemic episodes. To overcome these problems Space GlucoseControl was developed as a decision support system which helps to achieve safe and reliable blood glucose control in the desired ranges (4.4 - 6.1 mmol/l or 4.4 - 8.3 mmol/l).

The objective of this non-interventional study is to gain additional information on the performance of the Space GlucoseControl system for glycaemic control in ICU patients when used in routine clinical practice.

ELIGIBILITY:
Inclusion:

* Intensive care patients who require blood glucose control by intravenous application of insulin

Exclusion:

* All contraindication of intravenous insulin therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Blood glucose values: Percentage of time within the chosen glucose target range of 4.4 - 6.1 mmol/l or 4.4 - 8.3 mmol/l | From start of treatment to the last glucose measurement under treatment, typically up to 14 days.

SECONDARY OUTCOMES:
Frequency of hypoglycaemic episodes | From start of treatment to the last glucose measurement under treatment, typically up to 14 days.
Adherence to the advice of the Space GlucoseControl system | From start of treatment to the last glucose measurement under treatment, typically up to 14 days.
Blood glucose measurement interval | From start of treatment to the last glucose measurement under treatment, typically up to 14 days.

CONTACTS AND LOCATIONS:
Locations (17):
- Czechia (3):
  - Investigational Site, Hradec Králové
  - Investigational Site, Pilsen
  - Investigational sites, Prague
- Denmark (2):
  - Rigshospitalet Copenhagen, Copenhagen
  - Vejle Sygehus, Vejle
- Tartu University Hospital, Tartu, Estonia
- Germany (2):
  - Klinikum, Augsburg
  - Universitätsklinikum Leipzig, Leipzig
- Italy (2):
  - Investigational Site, Legnano
  - Investigational site, Siena
- Wroclaw Medical University, Wroclaw, Poland
- Hospital Sur,, Madrid, Spain
- Sweden (3):
  - Investigational Site, Jönköping
  - Investigational Site, Södertälje
  - Investigational Site, Stockholm
- United Kingdom (2):
  - West Suffolk Hospital, Bury Saint Edmonds
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Blaha J, Barteczko-Grajek B, Berezowicz P, Charvat J, Chvojka J, Grau T, Holmgren J, Jaschinski U, Kopecky P, Manak J, Moehl M, Paddle J, Pasculli M, Petersson J, Petros S, Radrizzani D, Singh V, Starkopf J. Space GlucoseControl system for blood glucose control in intensive care patients--a European multicentre observational study. BMC Anesthesiol. 2016 Jan 22;16:8. doi: 10.1186/s12871-016-0175-4. PMID 26801983